CLINICAL TRIAL: NCT02321917
Title: Coagulation, Inflammation and Cerebral Embolism Using a Rheoparin-coated Tubing System for Minimized Extracorporeal Circulation (MECC): Differences to the Conventional MECC System
Brief Title: Rheoparin-coated Tubing System for Minimized Extracorporeal Circulation (MECC)
Acronym: RheoMECC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 143/13
Record Dates: First submitted 2014-12-11; First posted 2014-12-22 (Estimated); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Extracorporeal Circulation; Inflammation; Blood Coagulation; Intracranial Embolism
MeSH Terms: conditions — Inflammation; Thrombosis; Intracranial Embolism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rheoparin coating (Active Comparator): MECC system with rheoparin coating
  Interventions: Device: MECC system with rheoparin coating
- No rheoparin coating (No Intervention): MECC system without rheoparin coating

INTERVENTIONS:
Device: MECC system with rheoparin coating — MECC system for extracorporeal circulation equipped with rheoparin coating.
  Arms: Rheoparin coating

SUMMARY:
In this study, the investigators would like to compare a heparin-coated tubing system for minimized extracorporeal circulation (MECC) with the conventional tubing system for MECC, which does not contain heparin coating. The MECC system has been used since 14 years in the investigators' hospital as an extracorporeal system to support circulation and provide oxygen to the tissues during coronary artery bypass grafting. Until today, the investigators performed more than 5000 MECC procedures in their department.

DETAILED DESCRIPTION:
Background

The investigators would like to investigate a new composition of their MECC system in patients receiving coronary artery bypass surgery. Normally, the MECC system induces complement system activation and coagulation cascade, which could have a negative impact on postoperative outcome. A tubing system containing heparin (rheoparin) could contribute to a better biocompatibility in terms of a diminished activation of inflammatory reactions and a reduction of cerebral embolic load, which is a regular issue during extracorporeal circulation due to formation of solid and gaseous microemboli in the tubing system.

Objective

The aim is to investigate biocompatibility (coagulation, inflammation) and influence on cerebral embolic load of the rheoparin-coated MECC system and to compare the results with the current MECC system containing a rheoparin-free tubing system.

Methods

Patients undergoing elective coronary artery surgery are randomized to receive extracorporeal circulation using the MECC system with or without rheoparin coating. All procedures are performed according to the institutional standards.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Elective cardiac surgery
* Coronary artery bypass grafting

Exclusion Criteria

* Re do
* Usage of antiplatelets, antithrombotic drugs
* Coagulopathy
* Persistent foramen ovale
* Infection
* Heparin-induced thrombocytopenia (HIT)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in coagulation / inflammation parameters at the post-operative phase | Perioperative period, 7 days
  Biocompatibility will be assessed by measuring different coagulatory and inflammatory parameters as determined in comparable studies. Especially, hte investigators assess in their central laboratory the thrombin-antithrombin complex and the d-dimer as measures of the activity of the coagulation/fibrinolysis system and furthermore the complement factors C3a-C5a, the interleukins IL 6, IL8, IL10, the tumor-necrosis factor alpha (TNF-alpha), platelet factor 4 and the syndecan-1 activity as an expression of the inflammatory response to the different coating used for minimized extracorporeal circulation system.

SECONDARY OUTCOMES:
Cerebral embolism | Perioperative period, 7 days
Mortality | At 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Carrel, MD, PhD, Principal Investigator — Dep. Cardiovascular Surgery
Locations (2):
- Switzerland (2):
  - Dep. Cardiovascular Surgery, Bern
  - Inselspital, University Hospital Bern, University of Bern, Bern